CLINICAL TRIAL: NCT06520007
Title: Comparison Between Continuous and Pulsed Oral Doxycycline Treatment Protocols for Refractory Meibomian Gland Dysfunction - 9 Months Follow-up Prospective Study
Brief Title: Comparison Between Continuous and Pulsed Oral Doxycycline Treatment Protocols for Refractory Meibomian Gland Dysfunction
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fogagnolo, Associate professor, University of Milan
Other Study IDs: CPDOXY1
Record Dates: First submitted 2024-07-13; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Meibomian Gland Dysfunction; Blepharitis; Doxycycline Adverse Reaction
Keywords: Meibomian gland dysfunction; Ocular surface disease; Doxycycline; Blepharitis
MeSH Terms: conditions — Meibomian Gland Dysfunction; Blepharitis | interventions — Doxycycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LCP - Low dose continuous protocol: Assumption of 50 mg of oral doxycycline per day for 3 months
  Interventions: Drug: Doxycyclin
- FPP - Full dose pulsed protocol: Assumption of 100 mg of oral doxycycline per day for 15 days per month (with a subsequent 15 days of washout) for 3 months
  Interventions: Drug: Doxycyclin

INTERVENTIONS:
Drug: Doxycyclin — The drug has been prescribed, as in normal clinical practice, with the National Healthcare System. Patients have been fully informed about interactions, toxicity and posology schedule.

SUMMARY:
The goal of this observational study (spontaneous, non-randomised, prospective cohort, phase IV) is to compare the efficacy and safety of two different oral doxycycline treatment protocols (LCP - Low dose continuous protocol & FPP - Full dose pulsed protocol) for meibomian gland dysfunction (MGD) in patients with refractory MGD (OSDI > 13 after at least 2 months treatment with warm compresses and lacrimal substitutes - first-line therapy). Systemic doxycycline doesn't have a standardized treatment protocol and this is why those patients are treated as in normal clinical practice. The main questions it aims to answer are:

Which treatment protocol has a greater impact on patient symptoms during the follow-up (OSDI score reduction)? Which treatment protocol has a greater impact on patient signs during the follow-up (TBUT and corneal staining variations)? Which treatment protocol is safer (in terms of adverse events rate)?

Participants will be visited every 3 months (V0-V1-V2-V3) with signs and symptoms assessment (TBUT, corneal staining, OSDI score) after being treated for 3 months with the assigned doxycycline treatment protocol (LCP or FPP).

DETAILED DESCRIPTION:
This spontaneous, prospective, non-randomized, parallel-group, phase IV study was conducted in compliance with the tenets of the Declaration of Helsinki.

All study participants were fully consented, and written informed consent was obtained.

This study included patients with refractory MGD. Refractory MGD is defined as symptomatic MGC (OSDI > 13 points) despite 2 months of first-line treatment with lacrimal substitutes 3 times per day and meibomian gland expression with warm compresses twice per day.

The study will consist of 3 visits: Baseline (day 0), Visit 2 (day 90 ± 5 - 3rd month), Visit 3 (day 180 ± 5 - 6 month). At each visit, patients will receive an OSDI questionnaire, NIBUT, type I Schirmer test and AS assessment, including TBUT, corneal staining (Oxford scale) At baseline, eligible patients will be enrolled and treated with the assigned protocol. The investigators will assign the protocol (non-randomized) in a 1:1 ratio.

At Visit 2, NIBUT, TBUT, Oxford scale and OSDI improvement will be evaluated compared with Visit 1. Patients will be carefully asked about their compliance with the treatment. Patients who interrupted the treatment for adverse events or low compliance (<75% of the protocol adherence) will exit the study and be excluded from the analysis.

At Visit 3, the study population will be evaluated as done in Visit 2

The protocols in the study are the following:

LCD (low-dose continuous protocol) - 50 mg of doxycycline for three months FPP ( Full-dose pulsed protocol) - 100 mg of doxycycline for the first 15 days of the month for three months.

The enrollment period will last about 6 months. Therefore, the study will end about 6 months after the last patient enrols.

ELIGIBILITY:
Inclusion criteria

* 18 years or older
* Provided written informed consent
* OSDI score of 13 or more at the baseline visit after at least two months of first-line therapy (artificial tears and warm compresses)
* Clinical diagnosis of MGD
* Type 1 Schirmer test > 10 mm
* No previous history of allergy or sensitivity to doxycycline,
* No use of additional topical or systemic antibiotics for the prior 2 months
* No use of topical anti-inflammatory agents (ex: corticosteroids or cyclosporine) for the prior 3 months.

Exclusion criteria

* Active ocular inflammation in either eye,
* Demodex blepharitis,
* Ocular surgery within the past 3 months of baseline examination,
* Structural ocular surface and eyelid abnormalities.
* Sjögren's syndrome
* Rheumatoid arthritis
* Other systemic diseases resulting in dry eye
* Known autoimmune disease
* Doxycycline allergy or sensitivity
* History of antibiotic therapy at any time within 2 months of the commencement of study
* Use of significant calcium supplementation or other medications that could interfere with doxycycline absorption (es: Iron supplementation)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory meibomian gland dysfunction (MGD). Refractory MGD is defined as symptomatic MGD (OSDI > 13 points) despite 2 months of first-line treatment with lacrimal substitutes 3 times per day and meibomian gland expression with warm compresses twice per day.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
OSDI score | Baseline - 3 months (90 days ± 5 days) - 6 months (180 days ± 5 days)
  Ocular Surface Disease Index

SECONDARY OUTCOMES:
TBUT | Baseline - 3 months (90 days ± 5 days) - 6 months (180 days ± 5 days)
  Tear break-up time
Corneal staining | Baseline - 3 months (90 days ± 5 days) - 6 months (180 days ± 5 days)
  Oxford scale has been use to assess corneal staining
Adverse events | From baseline up to the 3rd month
  Number of dropouts due to drug toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Santi Paolo e Carlo - Ospedale San Paolo, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT06520007/Prot_000.pdf